CLINICAL TRIAL: NCT05817747
Title: Strategic Use of Big Data in Spine Surgery - Testing a Digital Prediction of Outcome Tool in Clinical Praxis
Brief Title: Strategic Use of Big Data in Spine Surgery - Testing Digital Prediction of Outcome in Clinical Praxis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sahlgrenska University Hospital (Other)
Responsible Party: Principal Investigator, Catharina Parai, MD, PhD, Principal Investigator, Sahlgrenska University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022-2025
Record Dates: First submitted 2023-03-19; First posted 2023-04-18 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Constriction, Pathologic; Spine Degeneration; Surgery; Radiculopathy
Keywords: Spine; Cervical radiculopathy; Lumbar spinal stenosis; Surgery; Neck; Prognostic model; External validation
MeSH Terms: conditions — Constriction, Pathologic; Radiculopathy; Spinal Stenosis

STUDY DESIGN:
Intervention Model Description: On all participants the dialogue support tool will be used and will thereafter be put into either of two treatment-arms (surgical, or non-surgical treatment)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Surgery (Experimental): Participants will after the dialogue support tool has been undergo surgery.
  Interventions: Other: Dialogue support tool
- Non-surgery (Placebo Comparator): Participants will after the dialogue support tool has been used not undergo surgery.
  Interventions: Other: Dialogue support tool

INTERVENTIONS:
Other: Dialogue support tool — The dialogue support tool will be used as a support for the participant and surgeon to decide on which treatment arm is optimal for the participant.

SUMMARY:
The goal of this prospective, multicenter clinical trial is to determine if the use of the postoperative outcome prediction model the Dialogue Support tool can alter postoperative patient-reported outcome and satisfaction compared to current practice.

The main questions it aims to answer are:

* Does its use alter patient-reported outcome measured by general assessment regarding leg pain and Satisfaction in lumbar spinal stenosis?
* Does its use alter patient-reported outcome as measured by general assessment regarding arm pain and Satisfaction in cervical rhizopathy?
* How does the Quality of Life in patients - who after assessment by spinal surgeon do not proceed to surgery - compare with patients with the same baseline profile who did undergo surgery?

Eligible participants will be presented with their predicted postoperative outcome generated by the Dialogue Support tool, as an adjunct to the ordinary assessment by a spine surgeon.

Researchers will compare participants with a matched control group from the Swedish Spine Register ("Swespine") to see if the Dialogue Support tool can alter postoperative patient-reported outcome and satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Refered to a participating clinic regarding surgery for lumbar spinal stenosis or cervical radiculopathy
* 18 years of age or older
* Magnetic Resonance Imaging (MRT) examination within the last 12 months confirming the diagnosis, concurrent with symptoms described by the referring physician
* Giving informed consent

Exclusion Criteria:

* Another condition found to be the reason for the symptoms.
* Not giving informed consent
* Need for further investigation that prevents inclusion within one month of the doctor visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 900 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2027-03-01 (Estimated); Study Completion 2029-03-01 (Estimated)

PRIMARY OUTCOMES:
Global Assessment (GA) | One year post surgery
  A retrospective single-item question ("How is your back/leg or neck/arm pain today as compared to before the surgery?"), with six response options (not back/leg pain before surgery/completely gone/much improved/slightly improved/unchanged/worse).

SECONDARY OUTCOMES:
Oswestry Disability Index (ODI) | One year post surgery
  assesses the impact of lumbar pain on a patient´ physical function. It consists of ten questions concerning intensity of pain, ability to care for oneself, lifting, ability to walk, ability to sit, ability to walk, sexual function, social life, sleep quality and ability to travel. Min. value 0 points (no disability) and max. value 50 points (completely disabled).
Neck Disability index (NDI) | One year post surgery
  Used to assess the self-rated disability in patients with neck pain and consisting of ten questions scaled from 0-5 concerning pain-intensity, ability to care for oneself, lifting, reading, headache, concentration, working, driving, sleep and recreational activity
Euroqol-5-Dimensions quality of life questionnaire (EQ-5D) | One year post surgery
  Assess quality of life. It describes health in 5 dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. The five levels in each dimension are worded as (1) 'not /no problems', (2) 'slight problems', (3) 'moderate problems', (4) 'severe problems', and (5) 'unable to' (mobility, self-care, usual activities), 'extreme' (pain/depression), or 'extremely' (anxiety/depression).
Numeric Rating Scales for back/neck and leg/arm pain respectively (NRS) | One year post surgery
  The NRS is a common way of grading pain experience and is presented to the patient as a line with numbers from 0-10 and the patient is asked to grade their pain experience where zero is no pain and ten is maximal pain
Mortality | One year post surgery
  The number of participants that have died within one year of surgery

CONTACTS AND LOCATIONS:
Overall Officials: Catharina Parai, MD, PhD, Principal Investigator — Sahlgrenska University Hospital
Locations (10):
- Sweden (10):
  - Aleris Ortopedi Ängelholm, Ängelholm, Skåne County
  - Aleris Ortopedi Malmö, Malmo, Skåne County
  - Sahlgrenska University Hospital, Gothenburg, Västra Götaland County
  - Spine Center Göteborg, Gothenburg, Västra Götaland County
  - Ryggkirurgiskt Centrum, Stockholm
  - Spine Center Stockholm, Stockholm
  - Sundsvalls sjukhus, Sundsvall
  - Norrland University Hospital, Umeå
  - Uppsala University Hospital, Uppsala
  - Aleris Elisabethsjukhuset, Uppsala

REFERENCES:
- [Derived] Enger EB, Valentin-Askman L, Hagg O, Fritzell P, Parai C. The strategic use of Big Data - A study protocol for a multicenter clinical trial testing if the use of the Swespine Dialogue Support alter outcomes in degenerative spine surgery. BMC Musculoskelet Disord. 2024 Aug 21;25(1):654. doi: 10.1186/s12891-024-07714-5. PMID 39169349